CLINICAL TRIAL: NCT01252420
Title: Two Weeks of Low Molecular Weight Heparin for Distal Vein Thrombosis (TWISTER)
Brief Title: Two Weeks of Low Molecular Weight Heparin for Distal Vein Thrombosis
Acronym: TWISTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash Medical Centre (Other)
Collaborators: Southern Health, Victoria (Unknown); Eastern Health, Victoria (Unknown); Royal Adelaide Hospital, Adelaide (Unknown); Prince of Wales Hospital, Sydney (Other Government); Christchurch Hospital, NZ (Unknown); Auckland City Hospital (Other Government); North Shore Hospital, New Zealand (Other); Middlemore Hospital, New Zealand (Other)
Responsible Party: Huyen Tran, Monash Medical Centre, Southern Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDVTANZ
Record Dates: First submitted 2010-07-20; First posted 2010-12-03 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-07

CONDITIONS: Venous Thrombosis; Pulmonary Embolism
Keywords: Distal Vein Thrombosis; Proximal Vein Thrombosis; Pulmonary Embolism; Post-thrombotic syndrome; Limited duration treatment
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Postthrombotic Syndrome | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Enoxaparin — 1.5mg/kg daily for 2 weeks
  Other Names: Clexane

SUMMARY:
The purpose of this study is to determine whether a limited duration of treatment (two weeks of low molecular weight treatment) is a safe and effective treatment for distal deep vein thrombosis of the lower limb.

DETAILED DESCRIPTION:
Approximately 50% of symptomatic episodes of deep vein thrombosis (DVT) will be confined to the calf veins (distal DVT). The proportion of distal DVT that propagate to the proximal veins, increasing the risk of pulmonary embolism, is not known. The best treatment of isolated distal DVT is therefore controversial and options include no treatment, follow-up scanning and treatment of only those patients with thrombus propagating to proximal veins, and full anticoagulation for periods ranging from 2 weeks to 3 months.

There is good evidence that the 3-month thromboembolic risk in patients with a negative CUS that is limited to the proximal veins is low, in the order of 1%. Previous studies have demonstrated that patients treated with a short period of anticoagulation (4-6 weeks) have a low risk of developing recurrent DVT or PE. In addition, the specificity of CUS for distal DVT is lower than that for proximal DVT, increasing the proportion of false positive findings, making it likely that a proportion of patients diagnosed with distal DVT are treated unnecessarily, with the attendant risks of major and fatal haemorrhage.

The need for anticoagulation of patients with distal DVT to prevent recurrent DVT is therefore uncertain, however a survey of current practice suggested that most patients with this condition currently receive antithrombotic therapy. The impact of anticoagulation on initial patient symptoms, and the subsequent risk of the post-thrombotic syndrome are also unclear, and may be a possible alternative justification for antithrombotic therapy.

In this proposed multicentre, prospective, cohort study, we plan to determine if a shorter duration of anticoagulation (minimum 2 weeks) is a safe and effective treatment for isolated distal vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with acute symptomatic provoked or unprovoked distal vein thrombosis (axial or muscular veins but not involving trifurcation or distal popliteal vein)
* Absence of symptomatic pulmonary embolism

Exclusion Criteria:

* DVT involving trifurcation or more proximal leg veins on imaging
* Prior DVT
* Active malignancy ie present at time of diagnosis, or on treatment, or treatment completed within 3 months
* Ongoing risk factors for propagation e.g. immobility (>50% of day in bed or ≥72 hours), plaster cast or non-weight bearing
* Other indication for therapeutic anticoagulation (e.g. AF)
* Active gastro-oesophageal ulceration or bleeding
* Other high risk for bleeding (e.g. recent neurosurgery, vascular retinopathy, coagulopathy)
* Platelet count <80 x 109/L
* Renal impairment (CrCl <30ml/min) • Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Symptomatic recurrence of venous thrombosis (DVT, non fatal and fatal pulmonary embolism) within 3 months. | 3 months

SECONDARY OUTCOMES:
Asymptomatic proximal thrombus extension at 2 weeks | 2 weeks
Time course of symptom resolution and the proportion of patients with complete resolution at two weeks. | 2 weeks
  Time course of symptom resolution including time to complete resolution of symptoms, and the proportion of patients with complete resolution at two weeks.
All-cause mortality | 3 months
Post-thrombotic syndrome | 6 months
Predictors of recurrent or progressive DVT or new PE | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Huyen Tran, MBBs(Hons), MClin Epidem, Principal Investigator — Monash Medical Centre
Locations (4):
- Australia (3):
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Southern Health, Melbourne, Victoria
- Christchurch Hospital, Christchurch, Canterbury, New Zealand

REFERENCES:
- [Derived] Merriman E, Chunilal S, Brighton T, Chen V, McRae S, Ockelford P, Curnow J, Tran H, Chong B, Smith M, Royle G, Crowther H, Slocombe A, Tran H. Two Weeks of Low Molecular Weight Heparin for Isolated Symptomatic Distal Vein Thrombosis (TWISTER study). Thromb Res. 2021 Nov;207:33-39. doi: 10.1016/j.thromres.2021.09.004. Epub 2021 Sep 11. PMID 34530387